CLINICAL TRIAL: NCT00104481
Title: Cognitive Behavior Therapy for Smoking Cessation
Brief Title: Group Counseling for Smoking Cessation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: American University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R15CA077732-02A1 (NIH); 2R15CA077732-02A1 (NIH)
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2007-03

CONDITIONS: Smoking
Keywords: cognitive behavior therapy; coping; smoking cessation; acceptance; expectancies; quit smoking; quitting smoking
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: cognitive behavior therapy

SUMMARY:
The purpose of this study is to evaluate the effectiveness of group therapy for cigarette smoking cessation. The group meets for 8 sessions and includes education and group discussion about the effects of smoking and ways to cope with withdrawal symptoms and other challenges to maintaining abstinence. In one condition, the groups also learn techniques based on cognitive therapy, to help cope with negative feelings.

DETAILED DESCRIPTION:
The comparison condition is the same length as the cognitive behavior therapy condition but omits the cognitive restructuring component. In both conditions, smokers prepare for a quit date by using scheduled reduced smoking, which involves smoking on a set schedule that gradually reduces the number of cigarettes smoked. Post-treatment assessments occur one week after the end of treatment, and at 3-month followup.

Pre- and post-treatment assessments include measures of coping skills and emotional acceptance, as well as smoking rate.

ELIGIBILITY:
Inclusion Criteria:

* Regular daily smokers interested in quitting

Exclusion Criteria:

* Significant suicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-01; Study Completion 2007-08

PRIMARY OUTCOMES:
cigarette smoking abstinence

SECONDARY OUTCOMES:
cognitive coping skills
depressive symptoms
acceptance
distress tolerance

CONTACTS AND LOCATIONS:
Overall Officials: David A Haaga, Ph.D., Principal Investigator — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Haaga DA, Thorndike FP, Friedman-Wheeler DG, Pearlman MY, Wernicke RA. Cognitive coping skills and depression vulnerability among cigarette smokers. Addict Behav. 2004 Aug;29(6):1109-22. doi: 10.1016/j.addbeh.2004.03.026. PMID 15236811